CLINICAL TRIAL: NCT03523143
Title: The Effect of Early Screening and Intervention for Gestational Diabetes Mellitus on Pregnancy Outcomes: the TESGO Randomized Trial
Brief Title: The Effect of Early Screening and Intervention for Gestational Diabetes Mellitus on Pregnancy Outcomes
Acronym: TESGO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: At the interim analysis, the effect observed in this study was in the opposite direction in comparison to the original hypothesis. The three external experts decided that the trial should be stopped early according to pre-specified adaptation plans.
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201710072RINA
Record Dates: First submitted 2018-04-18; First posted 2018-05-14 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Pregnancy Complications; Gestational Diabetes Mellitus in Pregnancy
Keywords: early screening; early intervention; gestational diabetes mellitus; pregnancy outcomes; randomized controlled trial
MeSH Terms: conditions — Pregnancy Complications; Diabetes, Gestational | interventions — Methods

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early-screen Group (Experimental): The early screening group will be screened by a 75g 2-hour oral glucose tolerance test (OGTT) at 18-20 weeks of gestational age (GA). The time of early screening and intervention will be 6-8 weeks earlier than that of standard screening and intervention.
  Interventions: Other: early screening and intervention
- Standard-screen Group (Active Comparator): The standard screening group will be screened by a 75g 2-hour oral glucose tolerance test (OGTT) at 24-28 weeks of gestational age (GA). The time of standard screening and intervention will be 6-8 weeks later than that of early screening and intervention.
  Interventions: Other: standard screening and intervention

INTERVENTIONS:
Other: early screening and intervention — The early screening group will be screened by a 75g 2-hour oral glucose tolerance test (OGTT) at 18-20 weeks of gestational age (GA). Gestational diabetes mellitus (GDM) is diagnosed according to the IADPSG criteria. Subjects diagnosed with GDM will receive nutrition counseling, and lifestyle intervention. Pharmacologic therapies exclusively with human insulin or insulin analogues will be given when the target of glycemic control is not achieved within 4 weeks. The process of screening and intervention in the early screening group is all the same with that in the standard screening group. The only difference between two groups is the time of screening and intervention (18-20 weeks vs. 24-28 weeks of GA).
  Arms: Early-screen Group
Other: standard screening and intervention — The standard screening group will be screened by a 75g 2-hour oral glucose tolerance test (OGTT) at 24-28 weeks of gestational age (GA). Gestational diabetes mellitus (GDM) is diagnosed according to the International Association of Diabetes and Pregnancy Study Group (IADPSG) criteria, ie. if one of the plasma glucose levels at fasting, 1-hour, and 2-hour during OGTT is above 92 mg/dL, 180 mg/dL, and 153 mg/dL, respectively. Subjects diagnosed with GDM will receive nutrition counseling, and lifestyle intervention. Pharmacologic therapies exclusively with human insulin or insulin analogues will be given when the target of glycemic control is not achieved within 4 weeks.
  Arms: Standard-screen Group

SUMMARY:
Context: Women with gestational diabetes have excessive fetus growth weeks earlier than the screening period recommended currently, suggesting that earlier screening and intervention may improve pregnancy outcomes and the health of the offspring.

Objective: To determine if early screening and intervention could alter pregnancy outcomes, the incidence of maternal diabetes after delivery, and growth and development of the offspring, compared to the standard group.

Design, Setting, Participants: We will conduct a multi-center open-label randomized controlled trial in 2068 pregnant women, who deliver a singleton and who have not been diagnosed with overt diabetes mellitus at National Taiwan University Hospital (NTUH) and NTUH Hsinchu Branch from 2018 to 2020.

Interventions: Gestational diabetes mellitus (GDM) is diagnosed by a 75g 2-hour OGTT at 18-20 weeks of GA for the early-screening group and at 24-28 weeks for the standard-screening group. The diagnostic cutoffs are according to the IADPSG criteria. GDM is diagnosed if one of the plasma glucose levels at fasting, 1-hour, and 2-hour during OGTT is above 92 mg/dL, 180 mg/dL, or 153 mg/dL respectively. Subjects who are diagnosed with GDM receive lifestyle intervention and self-monitoring of blood glucose. Pharmacological therapies are given when the target of glycemic control is not achieved within 4-6 weeks.

Main Outcome Measure: The primary outcome is a composite measure of pregnancy outcomes, including primary CS, birth weight >90th percentile, neonatal hypoglycemia, cord serum C-peptide >90th percentile, pregnancy-induced hypertension, preeclampsia, and birth trauma. The primary outcome is measured within the entire period of perinatal and neonatal intensive-care units (NICU) stay for infants and the entire period of gestation for pregnant women after randomization.

Conclusion: This study will test our hypothesis that early screening and intervention of GDM improves pregnancy outcomes as compared to standard practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years old
2. First prenatal visit before 14 weeks of GA
3. Deliver a singleton at medical centers, including National Taiwan University Hospital (NTUH), and NTUH, Hsinchu Branch.

Exclusion Criteria:

1. Diagnosed with preexisting diabetes
2. Twin or multiple births pregnancy
3. Current exposure to steroids
4. Cannot tolerate an OGTT

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 967 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
TESGO composite outcome | The primary outcome is measured within the entire period of perinatal and NICU stay for infants and the entire period of gestation for pregnant women after randomization, an average of 10 months
  the occurrence rate of any of the following adverse outcome, including primary cesarean section (CS), birth weight >90th percentile, cord serum C-peptide ≥90th percentile, neonatal hypoglycemia, pregnancy-induced hypertension, preeclampsia, birth trauma, hypoglycemia, cord serum C-peptide >90th percentile, gestational hypertension, preeclampsia and birth trauma

SECONDARY OUTCOMES:
Preterm delivery | This secondary outcome is measured within the entire period of gestation for pregnant women after randomization, an average of 10 months
  the occurrence rate of preterm delivery
Jaundice | This secondary outcome is measured within the entire period of perinatal and NICU stay for infants, an average of 2 weeks
  the occurrence rate of newborns with jaundice
Admission to NICU | This secondary outcome is measured within the entire period of perinatal and NICU stay for infants, an average of 2 weeks
  the occurrence rate of newborns who need to be admitted to neonatal intensive care unit (NICU)
Fetal death or stillbirth | This secondary outcome is measured within the entire period of perinatal and NICU stay for infants and the entire period of gestation for pregnant women after randomization, an average of 10 months
  the occurrence rate of fetal death or stillbirth
Fetal growth during pregnancy | The secondary outcome is measured within the entire period of gestation for pregnant women after randomization, an average of 10 months
  measurement of fetal growth during pregnancy recorded by ultrasonography
Neonatal adiposity | The secondary outcome is measured within the entire period of perinatal and NICU stay for infants, an average of 2 weeks
  measurement of neonatal adiposity recorded by skinfold caliper
Maternal incident diabetes | This secondary outcome is measured during 3 years after delivery for eligible women
  the incidence of maternal diabetes after delivery
The growth and development of the offspring | This secondary outcome is measured during 3 years after delivery for eligible infants
  measurement of the growth and development of the offspring, including body height, body weight, head circumference, and records of any major disease

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Yuan Li, Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Internal Medicine, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tisi DK, Burns DH, Luskey GW, Koski KG. Fetal exposure to altered amniotic fluid glucose, insulin, and insulin-like growth factor-binding protein 1 occurs before screening for gestational diabetes mellitus. Diabetes Care. 2011 Jan;34(1):139-44. doi: 10.2337/dc10-0607. Epub 2010 Sep 20. PMID 20855548
- [Result] Qiu C, Vadachkoria S, Meryman L, Frederick IO, Williams MA. Maternal plasma concentrations of IGF-1, IGFBP-1, and C-peptide in early pregnancy and subsequent risk of gestational diabetes mellitus. Am J Obstet Gynecol. 2005 Nov;193(5):1691-7. doi: 10.1016/j.ajog.2005.04.015. PMID 16260212
- [Result] Asvold BO, Eskild A, Jenum PA, Vatten LJ. Maternal concentrations of insulin-like growth factor I and insulin-like growth factor binding protein 1 during pregnancy and birth weight of offspring. Am J Epidemiol. 2011 Jul 15;174(2):129-35. doi: 10.1093/aje/kwr067. Epub 2011 May 27. PMID 21622950
- [Result] Valensise H, Larciprete G, Vasapollo B, Novelli GP, Menghini S, di Pierro G, Arduini D. C-peptide and insulin levels at 24-30 weeks' gestation: an increased risk of adverse pregnancy outcomes? Eur J Obstet Gynecol Reprod Biol. 2002 Jul 10;103(2):130-5. doi: 10.1016/s0301-2115(02)00048-9. PMID 12069734
- [Result] Ning Y, Williams MA, Vadachkoria S, Muy-Rivera M, Frederick IO, Luthy DA. Maternal plasma concentrations of insulinlike growth factor-1 and insulinlike growth factor-binding protein-1 in early pregnancy and subsequent risk of preeclampsia. Clin Biochem. 2004 Nov;37(11):968-73. doi: 10.1016/j.clinbiochem.2004.07.009. PMID 15498523
- [Result] Lappas M. Insulin-like growth factor-binding protein 1 and 7 concentrations are lower in obese pregnant women, women with gestational diabetes and their fetuses. J Perinatol. 2015 Jan;35(1):32-8. doi: 10.1038/jp.2014.144. Epub 2014 Jul 31. PMID 25078866
- [Result] Sovio U, Murphy HR, Smith GC. Accelerated Fetal Growth Prior to Diagnosis of Gestational Diabetes Mellitus: A Prospective Cohort Study of Nulliparous Women. Diabetes Care. 2016 Jun;39(6):982-7. doi: 10.2337/dc16-0160. Epub 2016 Apr 7. PMID 27208333
- [Result] Gillman MW, Oakey H, Baghurst PA, Volkmer RE, Robinson JS, Crowther CA. Effect of treatment of gestational diabetes mellitus on obesity in the next generation. Diabetes Care. 2010 May;33(5):964-8. doi: 10.2337/dc09-1810. Epub 2010 Feb 11. PMID 20150300
- [Result] Landon MB, Rice MM, Varner MW, Casey BM, Reddy UM, Wapner RJ, Rouse DJ, Biggio JR Jr, Thorp JM, Chien EK, Saade G, Peaceman AM, Blackwell SC, VanDorsten JP; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units (MFMU) Network. Mild gestational diabetes mellitus and long-term child health. Diabetes Care. 2015 Mar;38(3):445-52. doi: 10.2337/dc14-2159. Epub 2014 Nov 20. PMID 25414152
- [Result] Gluckman PD, Hanson MA, Cooper C, Thornburg KL. Effect of in utero and early-life conditions on adult health and disease. N Engl J Med. 2008 Jul 3;359(1):61-73. doi: 10.1056/NEJMra0708473. No abstract available. PMID 18596274
- [Result] de Mello VD, Pulkkinen L, Lalli M, Kolehmainen M, Pihlajamaki J, Uusitupa M. DNA methylation in obesity and type 2 diabetes. Ann Med. 2014 May;46(3):103-13. doi: 10.3109/07853890.2013.857259. Epub 2014 Apr 30. PMID 24779963
- [Result] Waterland RA, Michels KB. Epigenetic epidemiology of the developmental origins hypothesis. Annu Rev Nutr. 2007;27:363-88. doi: 10.1146/annurev.nutr.27.061406.093705. PMID 17465856
- [Result] Lehnen H, Zechner U, Haaf T. Epigenetics of gestational diabetes mellitus and offspring health: the time for action is in early stages of life. Mol Hum Reprod. 2013 Jul;19(7):415-22. doi: 10.1093/molehr/gat020. Epub 2013 Mar 20. PMID 23515667
- [Result] International Association of Diabetes and Pregnancy Study Groups Consensus Panel; Metzger BE, Gabbe SG, Persson B, Buchanan TA, Catalano PA, Damm P, Dyer AR, Leiva Ad, Hod M, Kitzmiler JL, Lowe LP, McIntyre HD, Oats JJ, Omori Y, Schmidt MI. International association of diabetes and pregnancy study groups recommendations on the diagnosis and classification of hyperglycemia in pregnancy. Diabetes Care. 2010 Mar;33(3):676-82. doi: 10.2337/dc09-1848. No abstract available. PMID 20190296
- [Result] Metzger BE, Buchanan TA, Coustan DR, de Leiva A, Dunger DB, Hadden DR, Hod M, Kitzmiller JL, Kjos SL, Oats JN, Pettitt DJ, Sacks DA, Zoupas C. Summary and recommendations of the Fifth International Workshop-Conference on Gestational Diabetes Mellitus. Diabetes Care. 2007 Jul;30 Suppl 2:S251-60. doi: 10.2337/dc07-s225. No abstract available. PMID 17596481
- [Result] Workgroup on Hypoglycemia, American Diabetes Association. Defining and reporting hypoglycemia in diabetes: a report from the American Diabetes Association Workgroup on Hypoglycemia. Diabetes Care. 2005 May;28(5):1245-9. doi: 10.2337/diacare.28.5.1245. No abstract available. PMID 15855602
- [Result] Seaquist ER, Anderson J, Childs B, Cryer P, Dagogo-Jack S, Fish L, Heller SR, Rodriguez H, Rosenzweig J, Vigersky R. Hypoglycemia and diabetes: a report of a workgroup of the American Diabetes Association and the Endocrine Society. Diabetes Care. 2013 May;36(5):1384-95. doi: 10.2337/dc12-2480. Epub 2013 Apr 15. PMID 23589542